CLINICAL TRIAL: NCT03594617
Title: Improving Care and Preventing Maltreatment of Orphans: A Cluster-randomized Controlled Study With Caregivers
Brief Title: Improving Care and Preventing Maltreatment of Orphans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Collaborators: Bielefeld University (Other); Dar es Salaam University College of Education (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Elbert, Full Professor of Clinical Psychology and Behvavioral Neuroscience, University of Konstanz
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ICC-C-2018-Tanzania
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2019-09

CONDITIONS: Maltreatment, Child
MeSH Terms: interventions — Caregivers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICC-C (Experimental): Intervention: Interaction Competencies with children - for Caregivers (ICC-C) 11 days with 8 hours of training for caregivers. Core training components include caregiver-child interactions, maltreatment prevention, effective discipline strategies, child-centered institutional care, identifying and supporting burdened children and implementation of the training materials into the daily working
  Interventions: Behavioral: Interaction Competencies with Children - for Caregiver
- Control institutions (No Intervention): The control institutions do not receive any intervention.

INTERVENTIONS:
Behavioral: Interaction Competencies with Children - for Caregiver — Interaction Competencies with Children - for Caregiver (ICC-C) aims to reduce maltreatment and to improve care quality in institutional care facilities. Following the idea of a train-the-trainer approach, ICC-C is designed to be delivered by trained local facilitators. ICC-C is based on attachment, behavioral and social learning theories.
  The key principles are its feasibility in low-resource contexts, participatory approach, and practical orientation. ICC-C includes sessions on (a) caregiver-child interaction, (b) maltreatment prevention, (c) effective non-violent caregiving strategies, and (d) identifying and supporting burdened children.
  Arms: ICC-C

SUMMARY:
Sub-Saharan Africa, with more than 56 million orphans worldwide, is the most affected region in terms of orphans to be cared for (UNICEF, 2014). The recently developed preventative approach Interaction Competencies with Children - for Caregivers (ICC-C; Hecker, Mkinga, Ssenyonga, & Hermenau, 2017) trains the essential interaction skills in working with children. The focus here is on strengthening a warm, sensitive and reliable relationship between caregiver and child as well as on non-violent education strategies. In a first pilot study the feasibility of the approach icould be demonstrated (Hermenau, Kaltenbach, Mkinga, & Hecker, 2015).

The study applies a two-arm cluster-randomized controlled design. The participating institutions will be randomly divided into intervention and control bodies. The follow-up examination should take place three months after the intervention. All caregivers in facility (N = approx. 150) and 25 randomly selected children (age: 6-12) per facility (N = 200) will be included in this study.

DETAILED DESCRIPTION:
Sub-Saharan Africa, with more than 56 million orphans worldwide, is the most affected region in terms of orphans to be cared for (UNICEF, 2014). The few studies investigating children in African orphanages mostly showed inadequate care (Espié et al., 2011; Hermenau et al., 2011; Levin & Haines, 2007; Wolff & Fesseha, 1998, 1999). In addition to the lack of trained and competent caregivers, children are also confronted with violence and abuse in the orphanages themselves (Hermenau et al., 2011; SOS Children's Villages International & University of Bedfordshire, 2014). Abuse and neglect in orphanages, in addition to traumatisation, abuse and neglect in the families of origin, pose a considerable risk for the healthy development and mental health of children (Hermenau, Goessmann, Rygaard, Landolt, & Hecker, 2017). In addition to meeting basic needs (e. g. eating, drinking, basic medical care, etc.), sensitive and non-violent education in orphanages is crucial for the emotional and physical development of children. However, the focus of previous intervention studies has been on promoting a sensitive and reliable relationship between caregiver and child. Violence and maltreatment, on the other hand, received little attention (Hermenau et al., 2017).

The recently developed preventative approach Interaction Competencies with Children - for Caregivers (ICC-C; Hecker, Mkinga, Ssenyonga, & Hermenau, 2017) trains the essential interaction skills in working with children. The focus here is on strengthening a warm, sensitive and reliable relationship between caregiver and child as well as on non-violent education strategies. In a first pilot study the feasibility of the approach could be demonstrated (Hermenau, Kaltenbach, Mkinga, & Hecker, 2015).

The study applies a two-arm cluster-randomized controlled design and includes 20 to 25 orphanages. After an initial investigation, the participating institutions will be randomly divided into intervention and control bodies. The follow-up examination should take place three months after the intervention. In addition, feasibility data will be assessed in the intervention facilities only at the beginning and the end of the intervention. All caregivers in facility (N = approx. 150) and 10-15 randomly selected children (age: 6-12) per facility (N = 300) will be included in this study. Data of caregivers will be assessed with the help of self-administered questionnaires, whereas data of children will be assessed with structured interviews.

There is a clear and pressing humanitarian need for science to address the issue of care quality and maltreatment prevention in institutional care settings in a practical manner. Perhaps surprisingly in view of this, so far no evidenced-based prevention measures adapted for the limited resources in low-income countries have been developed and scientifically evaluated. This research project can address this need, with a scientifically rigorous evaluation of a violence and maltreatment prevention program that fosters the active involvement of local personnel and that considers the limited resources of school settings in low-income countries. Through these efforts this study may help more orphans to grow-up in a supportive atmosphere, maintaining their psychological well-being and improving their performance. This preventative program aims to make a significant impact on the psychological well-being of orphans in Tanzania.

ELIGIBILITY:
Inclusion Criteria for caregivers:

* Legal age
* Written informed consent

Inclusion Criteria for children:

* Between 6 and 12 years
* Written informed consent by head of institutional care facility & children oral assent

Exclusion Criteria for caregivers:

* Acute drug or alcohol intoxication
* Known psychiatric disorder

Exclusion Criteria for children:

- Known psychiatric disorder

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in caregivers' application of harsh discipline | The CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3-6 months after intervention)
  The Conflict Tactics Scale Parent-Child version (CTSPC) will assess caregiver's use of violent discipline measure against children in the child care institution. All items are rated on a 7-point Likert scale from never (0) to more than 20 times (25). The focus will be particularly on the subscales physical violence (13 items, potential range: 0 to 325 with higher scores indicating more violence) and emotional violence (5 items, potential range: 0-125, with higher scores indicating more violence).
Change in children's exposure to harsh discipline by caregivers | CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3-6 months after intervention)
  The Conflict Tactics Scale Parent-Child version (CTSPC) will assess the children's self-reported experiences of violent discipline in the child care institution. The focus will be particularly on the subscales physical violence (13 items, potential range: 0 to 325 with higher scores indicating more violence) and emotional violence (5 items, potential range: 0-125, with higher scores indicating more violence).

SECONDARY OUTCOMES:
Change in student's mental health | SDQ will be used at (baseline, prior to intervention) and T2 (follow-up, 3-6 months after intervention)
  Strength and Difficulties Questionnaire (SDQ) will assess children's internalizing and externalizing problems. The SDQ consists of five subscales of five items each, which are answered in three categories from "not true" (0), "somehow true" (1) to "certainly true" (2). The sum of all items except the ones from the prosocial behavior subscale represents atotal difficulty score (SDQ score; range 0-40, with a higher score indicating more problems). Values of 17 or higher on the SDQ score indicate severely elevated levels of mental health problems.
Change in caregiver's attitudes towards harsh discipline | The adapted version of CTSPC will be used at T 1 (baseline, prior to intervention) and T2 (follow-up, 3-6 months after intervention)
  Items of the Conflict Tactics Scale Parent-Child version (CTSPC) have been adapted to measure caregivers' and students' attitudes towards violent discipline methods in the child care institution. All items are rated on a 4-point Likert scale from never ok (0) to almost always ok (3). The focus will be particularly on the subscales physical violence (13 items, potential range: 0 to 39 with higher scores indicating more positive attitutudes towards violence) and emotional violence (5 items, potential range: 0-15, with higher scores indicating more positive attitudes towards violence).

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Hecker, PhD, Principal Investigator — Bielefeld University
Locations (1):
- Dar es Salaam University College of Education, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hecker T, Mkinga G, Hartmann E, Nkuba M, Hermenau K. Sustainability of effects and secondary long-term outcomes: One-year follow-up of a cluster-randomized controlled trial to prevent maltreatment in institutional care. PLOS Glob Public Health. 2022 May 20;2(5):e0000286. doi: 10.1371/journal.pgph.0000286. eCollection 2022. PMID 36962306
- [Derived] Hecker T, Mkinga G, Kirika A, Nkuba M, Preston J, Hermenau K. Preventing maltreatment in institutional care: A cluster-randomized controlled trial in East Africa. Prev Med Rep. 2021 Oct 9;24:101593. doi: 10.1016/j.pmedr.2021.101593. eCollection 2021 Dec. PMID 34976652